CLINICAL TRIAL: NCT06446713
Title: Proton Image-guided Radiation Assignment for Therapeutic Escalation Via Selection of Locally Advanced Head and Neck Cancer Patients
Brief Title: PIRATES: Image-guided Hyper-fractioned Dose-escalation With Proton Therapy for Head and Neck Cancer
Acronym: PIRATES
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18646
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer
Keywords: Proton therapy; Hyperfractionation; Dose-escalation; Image guidance therapy; Adaptive radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Single arm Bayesian Phase I intervention study
Masking Description: All participants receive the experimental treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Image guided hybrid hyper-fractioned dose escalation with proton therapy (Experimental)
  Interventions: Radiation: Image guided hybrid hyper-fractioned dose escalation with proton therapy

INTERVENTIONS:
Radiation: Image guided hybrid hyper-fractioned dose escalation with proton therapy — Radiation: Image-guided hybrid hyper-fractioned dose escalation with proton therapy
  The investigational radiation regime will be administered in a two-part schedule:
  * The first 4 weeks (i.e. first 20 fractions) of the radiation treatment of the pathological tumor will be according to the conventional clinical standard with proton therapy: 20x 2 Gy to the CTV70 and 20 x 1.55 Gy to the CTV54.
  * In week 4 (~ fraction 16) GTV80 will be determined on conventional weekly CT and additional MR imaging (conventional clinical protocol). Only this adapted tumor volume, the so-called GTV80, will receive the dose escalation (i.e., 80.5 Gy).
  * In the last 3 weeks (last 15 fractions) patients will be radiated twice per day (i.e. hyperfractionation). The GTV80, CTV70 and CTV54 will receive 1.55 Gy in the morning, and the GTV80 and CTV70 will receive additional dose in the afternoon.

SUMMARY:
In this study the safety & feasibility of image-guided mid-treatment hyper-fractioned dose-escalation with proton therapy will be assessed for the treatment of locally advanced HPV-negative squamous cell oropharyngeal cancer

DETAILED DESCRIPTION:
For this study, the investigators propose a novel design to safely achieve tumor radiation dose escalation with proton therapy plus standard-of-care concomitant chemotherapy. Through mid-treatment image guidance, the tumor boost dose is determined; subsequently, only that GTV boost will receive a total dose of 80 Gy through hybrid hyperfractionation. This refers to twice-daily radiation in the last 15 fraction days. The combination of boost dose hyperfractionation and proton therapy is anticipated to prevent critical normal tissue damage within both the high- and intermediate-dose regions. This novel treatment approach aims to minimize critical toxicities while improving locoregional control for head and neck cancer patients who are at a higher risk of disease relapse.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Biopsy proven diagnosis of squamous cell carcinoma originating in the oropharynx.
* Routine staging procedures, including CT of the head and neck region and chest, head and neck FDG-PET/CT and MRI (treatment planning allowed), and endoscopic evaluation when indicated.
* Negative for p16
* Locally advanced disease, specifically meeting all following criteria:

  * Stage III-IV
  * T-stage 2-4
  * All N-stages (N0-3)
  * M0
* Eligible for primary concurrent chemoradiation using conventionally fractionated radiotherapy 70 Gy combined with weekly cisplatin
* Eastern Cooperative Oncology Group (ECOG) performance score ≥2
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study; patients that:

* underwent definitive resection of their primary tumor or nodal disease, except for incisional or excisional biopsies.

received radiation therapy in the head and neck area in the past

* have no detectable tumor anymore at both the primary site and lymph nodes at week 4 in treatment, because there will not be a volume to boost.
* are unable or unwilling to give written, informed consent
* have contra-indications for chemotherapy. This is at the discretion of the treating medical oncologist.
* are unable to tolerate intravenous contrast for both CT and MRI, having an estimated GFR < 60 ml/min/1.73 m2 or any contraindications to gadolinium-based contrast agents.
* have any evidence of iron overload on pre-imaging laboratory studies.
* have other serious illnesses or medical conditions present at entry in the study, including (but not limited to): immunodeficiency virus (HIV) infection or other conditions of persistent immunodeficiency, neurologic or psychiatric disorders, active disseminated intravascular coagulation, unstable cardiac disease despite treatment or uncontrolled diabetes mellitus.
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility | Within 6 months after radiotherapy
  The number of dose limiting toxicity (DLT) events, defined as grade ≥4 mucositis, grade ≥4 ulceration, grade ≥4 dermatitis, grade ≥4 aspiration, grade ≥4 osteonecrosis and grade ≥3 myelopathy

SECONDARY OUTCOMES:
Completing radiotherapy regimen | End of radiotherapy
  Completion of treatment with a maximum of 2 fraction interruption
Completing chemotherapy regimen | End of chemotherapy
  Percentage of patients completing the complete chemotherapy regimen
Toxicity after chemoradiation | At 6 months after chemoradiation
  Rates of grade ≥3 mucositis, dermatitis, aspiration, dysphagia, hearing impaired, xerostomia, weight loss, trismus, hoarseness, oropharyngeal pain (according to CTCAEv5).
Tumor response rate | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  Preliminary tumor response rates measured on the standard follow-up MRI scan
Disease-free, overall survival and time-weighted locoregional control | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  Preliminary disease-free, overall survival and time-weighted locoregional control analyses

OTHER OUTCOMES:
Other physician rated toxicities | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  All other physician rated toxicities (CTCAEv5), including all grades
Patient-rated symptoms | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  Patient-rated symptoms (EORTC QLQ-H&N35)
Quality of life | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  Quality of life (EORTC QLQ-C30)
WHO performance | All SFP time points (baseline, weekly during RT, 6 weeks, 6, 12, 18, 24 months after treatment
  WHO performance

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided